CLINICAL TRIAL: NCT03725774
Title: The SUMAMOS EXCELENCIA Project: Assessment of Implementation of Best Practices in a National Health System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teresa Moreno Casbas (Other Government)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor-Investigator, Teresa Moreno Casbas, Head Of Nursing Research Unit, Instituto de Salud Carlos III
Organization: Instituto de Salud Carlos III (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI14CIII/00044
Record Dates: First submitted 2018-04-18; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-05

CONDITIONS: Age Problem
Keywords: pain; accidental falls; urinary incontinence; clinical audit
MeSH Terms: conditions — Pain; Urinary Incontinence | interventions — Hand Strength; Models, Biological

STUDY DESIGN:
Intervention Model Description: Uncontrolled before-and-after study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quasi-experimental uncontrolled, before-and-after (Experimental): The intervention will consist of the use of the GRIP (Getting Research into Practice) model and implementation of its strategies in clinical practice, according to the study unit in question and the scope of action
  Interventions: Other: GRIP (Getting Research into Practice) model

INTERVENTIONS:
Other: GRIP (Getting Research into Practice) model — The intervention will consist of the use of the GRIP (Getting Research into Practice) model and implementation of its strategies in clinical practice, according to the study unit in question and the scope of action.
  The GRIP model is a process of improvement by reference to a prior baseline clinical audit. It implies a local situation analysis, identifying the obstacles to improvements in clinical practice, and drawing up and implementing a plan of action for the purpose of improving adherence to pre-established criteria. The goal is to establish interprofessional processes within the teams, in order to: examine the obstacles that hinder the use of evidence in fostering best practices; and contribute to the development of implementation programmes for overcoming such obstacles.

SUMMARY:
There is a gap between research and clinical practice, leading to variability in decision-making. Clinical audits are an effective strategy for improving implementation of best practices. Quasi-experimental, multicentre, before-and-after. Primary-care and hospital-care units and associated socio-healthcare structures, and the patients attended at both. Implementation of evidence-based recommendations by application of the Getting Research into Practice model (process of improvement by reference to a prior baseline clinical audit. Data will be collected at baseline and, during the first year of follow up, at months (3, 6, 9,12)

DETAILED DESCRIPTION:
Aim: To assess the effectiveness of a model of implementation of evidence-based recommendations, in terms of patient outcomes and healthcare quality. Desing: Quasi-experimental, multicentre, before-and-after. Methods Primary-care and hospital-care units and associated socio-healthcare structures, and the patients attended at both. Intervention: Implementation of evidence-based recommendations by application of the Getting Research into Practice model (process of improvement by reference to a prior baseline clinical audit). Variables: Process and outcome criteria with respect to pain, urinary incontinence and fall prevention. Data will be collected at baseline and, during the first year of follow up, at months (3, 6, 9,12), with data on patients and indicators being drawn from clinical histories and records. Descriptive analysis, and comparison of the effectiveness of the intervention by means of inferential analysis and analysis of trends across follow-up. 95% confidence level. This project is funded by Spanish Strategic Health Action November 2014. Project duration 2015-2017.

ELIGIBILITY:
Inclusion Criteria:

* Unit-inclusion criteria. The study will cover all SNHS units and associated socio-healthcare structures which voluntarily adhere to the project and undertake to implement recommendations relating to pain, urinary incontinence and prevention falls.

For the purposes of this study, a "unit" is defined as any service, centre or institution that delivers health services to a homogeneous group of patients who share similar characteristics.

Patient-inclusion criteria. The study will include all patients attended at units participating in the study, who meet the following criteria, depending on the recommendations to be implemented at each unit:

* Pain: persons admitted to hospital centres who may potentially suffer from some type of pain. Patients will be classified according to whether they are adults or children (paediatric patients), and according to whether they experience chronic pain, acute postoperative pain, or acute pain due to other causes.
* Incontinence: community-dwelling or institutionalised persons prone to present with urinary incontinence. Patients will be classified according to whether they are 65 years of age or over.
* Falls: persons aged over 65 years who display one or more fall risk factors according to the assessment criteria established by the risk assessment instrument used.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence | 15 month
  Assessment of presence of urinary incontinence. Total number of patients in whom the presence of urinary incontinence has been initially assessed, and who are registered / Total number of patients discharged in the assessment period) * 100
Detection of pain, at admission | 15 month
  Total number of patients who have been assessed for the presence of pain and is registered / Total number of patients discharged during the measurement period) * 100 The assessment of the presence of pain will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of pain assessment with a Visual Analogic Scale (VAS; 10 cm, 0=no pain, 10=maximum pain) or Numerical rating scale (NRS; 0=no pain, 10 =worse pain), or the FLACC scale tool or paediatric patients,(Face, Leg, Activity, Cry, Consolability). Categories is scored from 0-2. Total scale: 0 is relaxed and comfortable, 1-2 Moderate discomfort, 3-6 Moderate pain and 7-10 Severe pain/discomfort f or PAINAD scale tool for patient with dementia. Measure breathing, negative vocalization, facial expression, body language and capacity for relief. Each item can get a maximum score of 2. The total scores can be from 0 (no pain) to 10 (maximum pain)
Risk of falls | 15 month
  Assessment of fall risk with a validated tool, at admission or onset of care.(Total number of patients to whom the risk of falls with a validated tool was initially assessed and registered / Total number of patients discharged during the measurement period) * 100 The assessment of fall risk in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of fall risk with a validated tools.Tools: Hendrich II Fall Risk Model, score: 0-16. Patient without risk (0), risk (1-4 points) and high risk (>5 points). H. Downton scale, score from 0 to 12. Patient without risk (0), low risk (1-2) and high risk (> 3 points). Morse Falls Scale, score from 0 to 150. Patient without risk (0-25), low risk (25-50) and high risk (> 50 points). Stratify or Stratify modified scale assesment includes five questions with dichotomous answer; obtaining two or more positive answer would classify the individual as a high risk patient to suffer a fall.

SECONDARY OUTCOMES:
Type of institution | 15 month
  hospital unit, primary care unit or socio-healthcare unit
Size of primary care unit | 15 month
  Population coverage will describe the size of primary care center.Number of patient assigned to the nurse
Size of socio-healthcare centres | 15 month
  The number of the beds assigned to the socio-healthcare
Size of hospital unit | 15 month
  number of beds assigned to the unit
nurse/patient ratio | 15 month
  number of patients per nurse
Age | 15 month
  Age of patients
Sex | 15 month
  Sex of patients
Reason for admission/consultation | 15 month
  Reason for admission/consultation of the patients. Reason for the patient to be admitted to the Hospital or to attend the consultation
Days of stay | 15month
  days of stay in the case of admissions
Impact of urinary incontinence | 15 month
  Impact of urinary incontinence.[Total number of patients with different urinary-incontinence impact levels 24 hours prior to assessment / Total number of patients attended during the data-collection period] * 100
Severity of incontinence | 15 month
  Patient education, urinary Incontinence management.[Total number of patients with different levels of severity of urinary incontinence 24 hours prior to assessment/ Total number of patients attended during the data-collection period] * 100
Type of urinary incontinence | 15 month
  Assessment of type of urinary incontinence. (Total number of incontinent patients with identification of type of incontinence, who are registered / Total number of incontinent patients) * 100
Patient education, urinary incontinence management. | 15 month
  (Number of patients with incontinence who receive (patients, family members or carers) incontinence management education at least once during the care process, and who are registered / Total number of patients with incontinence)*100
Urinary incontinence management | 15 month
  To establish and implement a comprehensive care plan to manage incontinence that includes: evaluation of results, believes, knowledge and level of comprehension of the patient, personal characteristics and incontinence characteristics. (Total number of incontinent patients that have a registered, multifactorial urinary incontinence management plan / Total number of incontinent patients) * 100
Pain at admission in paediatric patient | 15 month
  Detection of pain, at admission. (Total number of paediatric patients who have been assessed for the presence of pain and is registered / Total number of patients discharged during the measurement period) * 100 The assessment of the presence of pain will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of pain assessment with the FLACC scale tool (Face, Leg, Activity, Cry, Consolability). Categories is scored from 0-2. Total scale: 0 is relaxed and comfortable, 1-2 Moderate discomfort, 3-6 Moderate pain and 7-10 Severe pain/discomfort
Pain at admission in patient with dementia | 15 month
  Detection of pain, at admission. (Total number of patients with dementia who have been assessed for the presence of pain and is registered / Total number of patients discharged during the measurement period) * 100 The assessment of the presence of pain will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of pain assessment with the PAINAD scale (pain assesment in advanded dementia): tool for patient with dementia. Measure breathing, negative vocalization,facial expression, body language and capacity for relief. Each item can get a maximum score of 2. The total scores can be from 0 (no pain) to 10 (maximum pain)
Pain at admission in patient with mechanic ventilation | 15 month
  Detection of pain, at admission. (Total number of patients with mechanic ventilation who have been assessed for the presence of pain and is registered / Total number of patients discharged during the measurement period) * 100 The assessment of the presence of pain will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of pain assessment with the ESCID scale (Scale of Behavior Indicators of Pain). Mesaure: Facial expression, tranquility (movements), muscle tone, comfort and adaptation to mechanic ventilation. Each item is scored from 0 to 2; being 0 the minimum score and 10 the maximum.
Pain after a change in clinical status in adult patientfor pain | 15 month
  Detection of pain, after a change in clinical status. (Total number of adult patients who have been assessed for the presence of pain after change of clinical situation and is registered / Total number of adults patients discharged during the measurement period) * 100 The assessment of the presence of pain after a change in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of pain assessment with with a Visual Analogic Scale (VAS; 10 cm, 0=no pain, 10=maximum pain) or Numerical rating scale (NRS; 0=no pain, 10 =worse pain).
Pain after a change in clinical status in paediatric patient | 15 month
  Detection of pain, after a change in clinical status. (Total number of paediatric patients who have been assessed for the presence of pain after change of clinical situation and is registered / Total number of patients discharged during the measurement period) * 100 The assessment of the presence of pain after a change in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of pain assessment with a FLACC scale (Face, Leg, Activity, Cry, Consolability): tool for paediatric patient. Categories is scored from 0-2. Total scale: 0 is relaxed and comfortable, 1-2 Moderate discomfort, 3-6 Moderate pain and 7-10 Severe pain/discomfort
Pain after a change in clinical status in patient with dementia | 15 month
  Detection of pain, after a change in clinical status. (Total number of patients with dementia who have been assessed for the presence of pain after change of clinical situation and is registered / Total number of patients discharged during the measurement period) * 100 The assessment of the presence of pain after a change in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of pain assessment with a PAINAD scale (pain assesment in advanded dementia): tool for patient with dementia. Measure breathing, negative vocalization,facial expression, body language and capacity for relief. Each item can get a maximum score of 2. The total scores can be from 0 (no pain) to 10 (maximum pain)
Pain after a change in clinical status in patient with mechanic ventilation | 15 month
  Detection of pain, after a change in clinical status. (Total number of patients with dementia who have been assessed for the presence of pain after change of clinical situation and is registered / Total number of patients discharged during the measurement period) * 100 The assessment of the presence of pain after a change in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of pain assessment with a ESCID scale (Scale of Behavior Indicators of Pain). Tool for patient with mechanic ventilation. Mesaure: Facial expression, tranquility (movements), muscle tone, comfort and adaptation to mechanic ventilation. Each item is scored from 0 to 2; being 0 the minimum score and 10 the maximum.
Pain assessment | 15 month
  Pain assessment is defined as overall pain assessment in persons in whom the presence of pain has been detected, and identification of the type of pain (acute, chronic, nociceptive or neuropathic). (Total number of patients with identification of the type of pain and is registered / Total number of patients with pain) * 100 The assessment of the pain in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of the type of pain (acute, chronic, nociceptive or neuropathic)
Pain management | 15 month
  Establishing and implementing an overall pain management care plan for the patient which would include: evaluation of his/her outcomes, beliefs, knowledge, level of understanding and personal characteristics, and characteristics of the pain.(Total number of patients with pain who have a registered and multifactorial plan for pain management / Total number of patients with pain) * 100 The Pain management in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of evaluation of his/her outcomes, beliefs, knowledge, level of understanding and personal characteristics, and characteristics of the pain.
Patient education in pain | 15 month
  Patient education: collaborating with the patient in the identification of pain-control targets and appropriate strategies for an integrated approach to the care plan. (Number of patients with pain they receive (they, their family or caregivers) education about pain management at least once during the care process, and is registered / Total number of patients with pain) * 100
Intensity of Pain | 15 month
  ntensity of Pain assessment using a validated tool, for record-keeping purposes. [Total number of patients with pain intensity measurement / (Total number of patients attended during the data collection period] * 100
  The assessment of the intensity of pain in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of of the intensity of pain.
  The intensity of pain will be measured with different validated tools, according to whether the patient is an adult or paediatric, if he is conscious or not and if he has difficulty communicating.The tools are : Visual Analogic Scale (VAS), Numerical rating scale (NRS),FLACC Scale (Face, Leg, Activity, Cry, Consolability), PAINAD scale ( pain assesment in advanded dementia), ESCID scale (Scale of Behavior Indicators of PAin)
Maximum pain | 15 month
  Maximum score reported by a patient after pain-intensity assessment using a validated tool.
  The intensity of pain will be measured with different validated tools, according to whether the patient is an adult or paediatric, if he is conscious or not and if he has difficulty communicating.The tools are : Visual Analogic Scale (VAS), Numerical rating scale (NRS),FLACC Scale (Face, Leg, Activity, Cry, Consolability), PAINAD scale ( pain assesment in advanded dementia), ESCID scale (Scale of Behavior Indicators of PAin)
Risk after a fall | 15 month
  Assessment of fall risk with validated tool, after a fall. (Total number of patients who have been assessed the risk of falls with a validated tool after a fall and is registered / Total number of patients discharged in the measurement period) * 100 The assessment of fall risk after a fall in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of fall risk after a fall with a validated tools.Tools: Hendrich II Fall Risk Model, score: 0-16. Patient without risk (0), risk (1-4 points) and high risk (>5 points). H. Downton scale, score:0-12. Patient without risk (0), low risk (1-2) and high risk (> 3 points). Morse Falls Scale, score: 0-150. Patient without risk (0-25), low risk (25-50) and high risk (> 50 points). Stratify or Stratify modified scale assesment includes five questions with dichotomous answer; obtaining two or more positive answer would classify the individual as a high risk patient to suffer a fall.
Prevention of falls | 15 month
  Percentage of patients who are detected to be at risk using a fall-prevention plan or fall-injury reduction programme, based on a multifactorial approach, and are registered.
  The prevention of falls in clinical status will be measured in a dichotomous variable: Yes/No. For Yes, there must be registered evidence of are detected to be at risk using a fall-prevention plan or fall-injury reduction programme, based on a multifactorial approach, and are registered.
Use of restraints | 15 month
  Percentage of patients who are used restraints are physical, chemical or environmental measures used to control a person's physical or behavioural activity or a part of his/her body
Incidence of falls | 15 month
  Number of falls with or without injury among patients, per 1000 patients/day (acute care/rehabilitation/long stay) Total number of falls with or without injury, per 1000 patients (primary care)
Falls that cause injury | 15 month
  Percentage of falls resulting in mild, moderate, severe injury or death, according to the WHO classification.
  Injury is defined as bodily harm suffered as a consequence of a fall.

CONTACTS AND LOCATIONS:
Overall Officials: TERESA MORENO CASBAS, DOCTOR, Study Director — Instituto de Salud Carlos III; ESTHER GONZALEZ MARIA, DOCTOR, Study Chair — Instituto de Salud Carlos III; ISABEL ORTS CORTÉS, DOCTOR, Study Chair — UNIVERSIDAD DE ALICANTE; CLARA SANCHEZ PABLO, RN, Study Chair — Instituto de Salud Carlos III

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albornos-Muñoz, L., González-María, E., Moreno-Casbas, T. (2015). Implantación de Guías de Buenas Prácticas en España. Programa de Centros Comprometidos con la Excelencia en Cuidados® (Best Practice Guidelines Implementation in Spain. Best Practice Spotlight Organizations ® Programme). MedUNAB, 17(3), pp. 163-69.
- [Result] Baker R, Camosso-Stefinovic J, Gillies C, Shaw EJ, Cheater F, Flottorp S, Robertson N. Tailored interventions to overcome identified barriers to change: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD005470. doi: 10.1002/14651858.CD005470.pub2. PMID 20238340
- [Result] Bauer MS, Damschroder L, Hagedorn H, Smith J, Kilbourne AM. An introduction to implementation science for the non-specialist. BMC Psychol. 2015 Sep 16;3(1):32. doi: 10.1186/s40359-015-0089-9. PMID 26376626
- [Result] Bero LA, Grilli R, Grimshaw JM, Harvey E, Oxman AD, Thomson MA. Closing the gap between research and practice: an overview of systematic reviews of interventions to promote the implementation of research findings. The Cochrane Effective Practice and Organization of Care Review Group. BMJ. 1998 Aug 15;317(7156):465-8. doi: 10.1136/bmj.317.7156.465. No abstract available. PMID 9703533
- [Result] Bornbaum CC, Kornas K, Peirson L, Rosella LC. Exploring the function and effectiveness of knowledge brokers as facilitators of knowledge translation in health-related settings: a systematic review and thematic analysis. Implement Sci. 2015 Nov 20;10:162. doi: 10.1186/s13012-015-0351-9. PMID 26589972
- [Result] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Result] Davies B, Edwards N, Ploeg J, Virani T. Insights about the process and impact of implementing nursing guidelines on delivery of care in hospitals and community settings. BMC Health Serv Res. 2008 Feb 2;8:29. doi: 10.1186/1472-6963-8-29. PMID 18241349
- [Result] Dobbins M, Cockerill R, Barnsley J, Ciliska D. Factors of the innovation, organization, environment, and individual that predict the influence five systematic reviews had on public health decisions. Int J Technol Assess Health Care. 2001 Fall;17(4):467-78. PMID 11758291
- [Result] Estabrooks CA. The conceptual structure of research utilization. Res Nurs Health. 1999 Jun;22(3):203-16. doi: 10.1002/(sici)1098-240x(199906)22:33.0.co;2-9. PMID 10344701
- [Result] Flodgren G, Deane K, Dickinson HO, Kirk S, Alberti H, Beyer FR, Brown JG, Penney TL, Summerbell CD, Eccles MP. Interventions to change the behaviour of health professionals and the organisation of care to promote weight reduction in overweight and obese people. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD000984. doi: 10.1002/14651858.CD000984.pub2. PMID 20238311
- [Result] Forbes A, Griffiths P. Methodological strategies for the identification and synthesis of 'evidence' to support decision-making in relation to complex healthcare systems and practices. Nurs Inq. 2002 Sep;9(3):141-55. doi: 10.1046/j.1440-1800.2002.00146.x. PMID 12199878
- [Result] Mc Goldrick EL, Crawford T, Brown JA, Groom KM, Crowther CA. Identifying the barriers and enablers in the implementation of the New Zealand and Australian Antenatal Corticosteroid Clinical Practice Guidelines. BMC Health Serv Res. 2016 Oct 28;16(1):617. doi: 10.1186/s12913-016-1858-8. PMID 27793150
- [Result] Graham ID, Logan J, Harrison MB, Straus SE, Tetroe J, Caswell W, Robinson N. Lost in knowledge translation: time for a map? J Contin Educ Health Prof. 2006 Winter;26(1):13-24. doi: 10.1002/chp.47. PMID 16557505
- [Result] Grimshaw JM, Russell IT. Effect of clinical guidelines on medical practice: a systematic review of rigorous evaluations. Lancet. 1993 Nov 27;342(8883):1317-22. doi: 10.1016/0140-6736(93)92244-n. PMID 7901634
- [Result] Grimshaw J, Eccles M, Thomas R, MacLennan G, Ramsay C, Fraser C, Vale L. Toward evidence-based quality improvement. Evidence (and its limitations) of the effectiveness of guideline dissemination and implementation strategies 1966-1998. J Gen Intern Med. 2006 Feb;21 Suppl 2(Suppl 2):S14-20. doi: 10.1111/j.1525-1497.2006.00357.x. PMID 16637955
- [Result] Grimshaw JM, Eccles MP, Lavis JN, Hill SJ, Squires JE. Knowledge translation of research findings. Implement Sci. 2012 May 31;7:50. doi: 10.1186/1748-5908-7-50. PMID 22651257
- [Result] Grimshaw JM, Thomas RE, MacLennan G, Fraser C, Ramsay CR, Vale L, Whitty P, Eccles MP, Matowe L, Shirran L, Wensing M, Dijkstra R, Donaldson C. Effectiveness and efficiency of guideline dissemination and implementation strategies. Health Technol Assess. 2004 Feb;8(6):iii-iv, 1-72. doi: 10.3310/hta8060. PMID 14960256
- [Result] Grol R, Grimshaw J. From best evidence to best practice: effective implementation of change in patients' care. Lancet. 2003 Oct 11;362(9391):1225-30. doi: 10.1016/S0140-6736(03)14546-1. PMID 14568747
- [Result] Hunskaar S, Lose G, Sykes D, Voss S. The prevalence of urinary incontinence in women in four European countries. BJU Int. 2004 Feb;93(3):324-30. doi: 10.1111/j.1464-410x.2003.04609.x. PMID 14764130
- [Result] Kajermo KN, Bostrom AM, Thompson DS, Hutchinson AM, Estabrooks CA, Wallin L. The BARRIERS scale -- the barriers to research utilization scale: A systematic review. Implement Sci. 2010 Apr 26;5:32. doi: 10.1186/1748-5908-5-32. PMID 20420696
- [Result] Kitson A, Ahmed LB, Harvey G, Seers K, Thompson DR. From research to practice: one organizational model for promoting research-based practice. J Adv Nurs. 1996 Mar;23(3):430-40. doi: 10.1111/j.1365-2648.1996.tb00003.x. PMID 8655816
- [Result] Kreindler SA. What if implementation is not the problem? Exploring the missing links between knowledge and action. Int J Health Plann Manage. 2016 Apr;31(2):208-26. doi: 10.1002/hpm.2277. Epub 2014 Nov 25. PMID 25424863
- [Result] Langley PC, Ruiz-Iban MA, Molina JT, De Andres J, Castellon JR. The prevalence, correlates and treatment of pain in Spain. J Med Econ. 2011;14(3):367-80. doi: 10.3111/13696998.2011.583303. Epub 2011 May 17. PMID 21574899
- [Result] Meijers JM, Janssen MA, Cummings GG, Wallin L, Estabrooks CA, Y G Halfens R. Assessing the relationships between contextual factors and research utilization in nursing: systematic literature review. J Adv Nurs. 2006 Sep;55(5):622-35. doi: 10.1111/j.1365-2648.2006.03954.x. PMID 16907795
- [Result] Milner M, Estabrooks CA, Myrick F. Research utilization and clinical nurse educators: A systematic review. J Eval Clin Pract. 2006 Dec;12(6):639-55. doi: 10.1111/j.1365-2753.2006.00632.x. PMID 17100863
- [Result] Pallen N, Timmins F. Research-based practice: myth or reality? A review of the barriers affecting research utilisation in practice. Nurse Educ Pract. 2002 Jun;2(2):99-108. doi: 10.1054/nepr.2002.0058. PMID 19036286
- [Result] Pearson A. Getting research into practice. Int J Nurs Pract. 2004 Oct;10(5):197-8. doi: 10.1111/j.1440-172X.2004.00486.x. No abstract available. PMID 15461688
- [Result] Rycroft-Malone J. Theory and knowledge translation: setting some coordinates. Nurs Res. 2007 Jul-Aug;56(4 Suppl):S78-85. doi: 10.1097/01.NNR.0000280631.48407.9b. PMID 17625479
- [Result] Ruzafa-Martinez M, Gonzalez-Maria E, Moreno-Casbas T, del Rio Faes C, Albornos-Munoz L, Escandell-Garcia C. [The Spanish best practice guidelines implementation project 2011-2016]. Enferm Clin. 2011 Sep-Oct;21(5):275-83. doi: 10.1016/j.enfcli.2011.07.013. Epub 2011 Sep 15. Spanish. PMID 21924654
- [Result] Sackett DL, Rosenberg WM, Gray JA, Haynes RB, Richardson WS. Evidence based medicine: what it is and what it isn't. BMJ. 1996 Jan 13;312(7023):71-2. doi: 10.1136/bmj.312.7023.71. No abstract available. PMID 8555924
- [Result] Schuster MA, McGlynn EA, Brook RH. How good is the quality of health care in the United States? Milbank Q. 1998;76(4):517-63, 509. doi: 10.1111/1468-0009.00105. PMID 9879302
- [Result] Shaneyfelt TM, Mayo-Smith MF, Rothwangl J. Are guidelines following guidelines? The methodological quality of clinical practice guidelines in the peer-reviewed medical literature. JAMA. 1999 May 26;281(20):1900-5. doi: 10.1001/jama.281.20.1900. PMID 10349893
- [Result] Squires JE, Estabrooks CA, Gustavsson P, Wallin L. Individual determinants of research utilization by nurses: a systematic review update. Implement Sci. 2011 Jan 5;6:1. doi: 10.1186/1748-5908-6-1. PMID 21208425
- [Result] Stergiou-Kita M. Implementing Clinical Practice Guidelines in occupational therapy practice: recommendations from the research evidence. Aust Occup Ther J. 2010 Apr;57(2):76-87. doi: 10.1111/j.1440-1630.2009.00842.x. PMID 20854572
- [Result] Thomas L, Cullum N, McColl E, Rousseau N, Soutter J, Steen N. Guidelines in professions allied to medicine. Cochrane Database Syst Rev. 2000;(2):CD000349. doi: 10.1002/14651858.CD000349. PMID 10796531
- [Derived] Escobar-Aguilar G, Moreno-Casbas MT, Gonzalez-Maria E, Martinez-Gimeno ML, Sanchez-Pablo C, Orts-Cortes I. The SUMAMOS EXCELENCIA Project. J Adv Nurs. 2019 Jul;75(7):1575-1584. doi: 10.1111/jan.13988. Epub 2019 Apr 2. PMID 30816569